CLINICAL TRIAL: NCT02689765
Title: Effect of Anthocyanins on Metabolic Profiles in Subjects With Pre-diabetes: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Anthocyanins on Metabolic Profiles in Subjects With Pre-diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, LiPing Yang, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20151218
Record Dates: First submitted 2016-02-19; First posted 2016-02-24 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Insulin Resistance; Glucose Metabolism Disorders; Type 2 Diabetes; Lipid Metabolism Disorders
MeSH Terms: conditions — Insulin Resistance; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Lipid Metabolism Disorders | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anthocyanins (Experimental): Volunteers will be randomised double blinded into 'Anthocyanins' groups(n=60 per group)and given twice daily two capsules of either 80 grams of Anthocyanins, which corresponds a mixture of fresh blue berries and blackcurrants.The total duration of this trial was 24wk.
  Interventions: Dietary Supplement: Anthocyanins
- Control (Placebo Comparator): A daily intake of 320mg Placebo to instead of treatment of Anthocyanins.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Anthocyanins — Anthocyanins capsules, which comprises different natural Anthocyanins purified from bilberries and blackcurrants
  Other Names: Medox
  Arms: Anthocyanins
Dietary Supplement: Placebo — Placebo capsules is identically packaged.
  Arms: Control

SUMMARY:
Metabolic problems represent one of the major health concerns which are attractive for being addressed by nutritional interventions, as these are directly connected to dietary habits.Anthocyans possess cardiovascular disease prevention, obesity control, and diabetes alleviation properties, but association between anthocyans and prediabetes need to be more firmly understood and established from robust clinical data. However, there is little human research that has reported on the efficacy of increased anthocyans bioactive consumption on insulin sensitivity in pre-diabetes.

DETAILED DESCRIPTION:
The investigators plan to conduct a randomized double-blind, placebo-controlled trial to characterize the potential effects of anthocyans, purified from bilberries and blackcurrants, on metabolic abnormalities commonly associated with type 2 pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* FPG 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L) (IFG) OR 2-h plasma glucose in the 75gOGTT 140 mg/dL (7.8 mmol/L) to 199 mg/dL (11.0 mmol/L)(IGT) OR HbA1C 5.7-6.4%.
* Newly diagnosed T2DM who exceed the upper limit of the range but has not yet accepted hypoglycemic therapy.

Exclusion Criteria:

Patients with cardiac, renal, or hepatic diseases or with hyperthyroidism or who had concomitant infections, or who use of anti-diabetic drug or potential affect plasma glucose drugs, pregnant and breast-feeding women, and with polycystic ovarian syndrome.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in fasting glucose and HbA1C | 12 weeks

SECONDARY OUTCOMES:
The area under the curves for Glucose,insulin and C peptide releasing test(fasting and post 75g oral glucose tolerance test) | 12 weeks
Lipids | 12 weeks
  Total cholesterol,Triglycerides,HDL cholesterol,LDL cholesterol,Apolipoprotein A-I ,Apolipoprotein B
Calculated pancreatic β-cell function and insulin resistance | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Baiyun Street Hospital,Yuexiu District, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang L, Liu Z, Ling W, Wang L, Wang C, Ma J, Peng X, Chen J. Effect of Anthocyanins Supplementation on Serum IGFBP-4 Fragments and Glycemic Control in Patients with Fasting Hyperglycemia: A Randomized Controlled Trial. Diabetes Metab Syndr Obes. 2020 Sep 28;13:3395-3404. doi: 10.2147/DMSO.S266751. eCollection 2020. PMID 33061500
- [Derived] Yang L, Ling W, Qiu Y, Liu Y, Wang L, Yang J, Wang C, Ma J. Anthocyanins increase serum adiponectin in newly diagnosed diabetes but not in prediabetes: a randomized controlled trial. Nutr Metab (Lond). 2020 Sep 21;17:78. doi: 10.1186/s12986-020-00498-0. eCollection 2020. PMID 32973912
- [Derived] Yang L, Qiu Y, Ling W, Liu Z, Yang L, Wang C, Peng X, Wang L, Chen J. Anthocyanins regulate serum adipsin and visfatin in patients with prediabetes or newly diagnosed diabetes: a randomized controlled trial. Eur J Nutr. 2021 Jun;60(4):1935-1944. doi: 10.1007/s00394-020-02379-x. Epub 2020 Sep 15. PMID 32930848
- See also: The effects of purified anthocyanins on dyslipidemia, oxidative status, and insulin sensitivity in patients with type 2 diabetes. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Purified+anthocyanin+supplementation+reduces+dyslipidemia%2C+enhances+antioxidant+capacity%2C+and+prevents+insulin+resistance+in+diabetic+patients
- See also: The effects of anthocyanin supplementation on insulin resistance and liver injury biomarkers in patients with NAFLD. — http://www.ncbi.nlm.nih.gov/pubmed/?term=A+CONSORT-compliant%2C+randomized%2C+double-blind%2C+placebo-controlled+pilot+trial+of+purified+anthocyanin+in+patients+with+nonalcoholic+fatty+liver+disease
- See also: The supplementation of an anthocyanin mixture to hypercholesterolemic subjects for 24 weeks reduced serum levels of CRP, VCAM-1 and IL-1b, which involved the improvement of the lipid profile — http://www.ncbi.nlm.nih.gov/pubmed/?term=Anti-inflammatory+effect+of+purified+dietary+anthocyanin+in+adults+with+hypercholesterolemia%3A+a+randomized+controlled+trial